CLINICAL TRIAL: NCT00382720
Title: A Randomized Phase II Study of Docetaxel in Combination With Oxaliplatin With or Without 5-FU or Capecitabine in Metastatic or Locally Recurrent Gastric Cancer Previously Untreated With Chemotherapy for Advanced Disease
Brief Title: Docetaxel and Oxaliplatin in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCOX_C_00082; EudraCT # : 2005-005464-92
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Fluorouracil; Capecitabine

ARMS (3):
- TE (Taxotere and Eloxatin) (Experimental): Docetaxel (Taxotere) in combination with Oxaliplatin (Eloxatin). Each chemotherapy cycle was repeated every 21 days.
  Participants received either the optimal or non-optimal dose for Taxotere and Eloxatin. Participants who received the optimal dose for Taxotere and Eloxatin were analyzed in this study.
  Interventions: Drug: Docetaxel + Oxaliplatin
- TEF (Taxotere, Eloxatin and 5-FU) (Experimental): Docetaxel (Taxotere) in combination with Oxaliplatin (Eloxatin) and 5-FU (5-Fluorouracil). Each chemotherapy cycle was repeated every 14 days.
  Participants received either the optimal or non-optimal dose for Taxotere, Eloxatin and 5-FU. Participants who received the optimal dose for Taxotere, Eloxatin and 5-FU were analyzed in this study.
  Interventions: Drug: Docetaxel + Oxaliplatin + 5-FU
- TEX (Taxotere, Eloxatin and Xeloda) (Experimental): Docetaxel (Taxotere) in combination with Oxaliplatin (Eloxatin) and capecitabine (Xeloda). Each chemotherapy cycle was repeated every 21 days.
  Participants received either the optimal or non-optimal dose for Taxotere, Eloxatin and Xeloda. Participants who received the optimal dose for Taxotere, Eloxatin and Xeloda were analyzed in this study.
  Interventions: Drug: Docetaxel + Oxaliplatin + Capecitabine

INTERVENTIONS:
Drug: Docetaxel + Oxaliplatin — Dose level 1 (non-optimal dose):
  Docetaxel 75 mg/m² as an 1-hour intravenous (IV) infusion on day 1 followed by Oxaliplatin 100 mg/m² as a two to six-hour IV infusion on day 1
  Dose level 2 (optimal dose):
  Docetaxel 75 mg/m² as an 1-hour IV infusion on day 1 followed by Oxaliplatin 130 mg/m² as a two to six-hour IV infusion on day 1
  Arms: TE (Taxotere and Eloxatin)
Drug: Docetaxel + Oxaliplatin + 5-FU — Dose level 1 (non-optimal dose):
  Docetaxel 40 mg/m² as a 1-hour intravenous (IV) infusion day 1; Oxaliplatin 85 mg/m² simultaneously with folinic acid 400 mg/m² as a 2-hour IV infusion, followed by 5-FU 2400 mg/m2 as a 46-hour continuous infusion day 1.
  Dose level 2 (optimal dose):
  Docetaxel 50 mg/m² as a 1-hour IV infusion day 1; Oxaliplatin 85 mg/m² simultaneously with folinic acid 400 mg/m² as a 2-hour IV infusion, followed by 5-FU 2400 mg/m² as a 46-hour continuous infusion day 1.
  Arms: TEF (Taxotere, Eloxatin and 5-FU)
Drug: Docetaxel + Oxaliplatin + Capecitabine — Dose level 1 (optimal dose):
  Docetaxel 50 mg/m² as a 1-hour intravenous (IV) infusion on day 1, Oxaliplatin 100 mg/m² as a two to six-hour IV infusion on day 1, Capecitabine 625 mg/m2 two times a day continuously.
  Dose level 2 (non-optimal dose):
  Docetaxel 65 mg/m² as a 1-hour IV infusion on day 1, Oxaliplatin 100 mg/m² as a two to six-hour IV infusion on day 1, Capecitabine 625 mg/m² two times a day continuously.
  Arms: TEX (Taxotere, Eloxatin and Xeloda)

SUMMARY:
This phase II study addressed the use of docetaxel in combination with oxaliplatin with or without 5-FU or capecitabine in metastatic or locally recurrent gastric cancer previously untreated with chemotherapy for advanced disease. Prior to this study a pilot phase I (part I) determined the optimal dose by assessing the safety and tolerability of 2 dose levels in each arm. The optimal dose was administered in the Part II study. Participants who received the optimal dose in each treatment arm in Part I were included in the Part II analysis population.

Primary objective:

* To assess the time to progression (TTP) of Docetaxel in combination with Oxaliplatin with or without 5-Fluorouracil (5-FU) or Capecitabine in metastatic or locally recurrent gastric cancer previously untreated with chemotherapy for advanced disease (part II).

Secondary objectives:

* To establish the safety profile.
* To assess the Overall Response Rate (ORR) based on the World Health Organization (WHO) criteria
* To assess the Overall Survival (OS)

DETAILED DESCRIPTION:
The purpose of this study (Part II) was to evaluate the time to progression in the 3 arms at an optimal dose level of docetaxel and oxaliplatin defined during a prior pilot (Part I) phase study. The estimated duration of treatment was to be 6 months. Treatment was to be administered up to progression, unacceptable toxicities, or withdrawal of consent. The reason and date of removal of all participants was documented on the case report form.

Participants who ended treatment but had not yet progressed (e.g. unacceptable toxicities or withdrawal of consent) were be followed every 8 weeks with a complete tumor assessment until documented progression or further anti-tumor therapy. Then, they would be followed every 3 months after progression for survival status; date of death or progression were reported. Participants who ended treatment for progression, were to be followed every 3 months until death. Date of death was reported. The planned duration of the study was 30 months.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven gastric adenocarcinoma, including adenocarcinoma of the gastro-oesophageal junction
* Metastatic or locally recurrent disease
* Prior adjuvant (and/or neo-adjuvant) chemotherapy with 5-Fluorouracil, Cisplatin, epirubicin is allowed provided that the patient has relapsed > 12 months after the end of the chemotherapy
* Performance status Karnofsky index > 70
* Hematology within 7 days before randomization:Hemoglobin ≥10g/dl, Absolute Neutrophil Count ≥2.0 10^9/L, platelets ≥100 x 10^9/L
* Blood chemistry within 7 days before randomization:Total bilirubin ≤1x Upper Normal Limit(UNL), Aspartate Aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase SGOT) and Alanine Aminotransferase (ALT)Serum Glutamate Pyruvate Transaminase(SGPT) ≤2.5xUNL, alkaline phosphatase ≤ 5x UNL, provided that AST or ALT > 1.5 x UNL is not associated with alkaline phosphatase > 2.5 x UNL; creatinine ≤1.25x UNL or 1.25x UNL < creatinine ≤1.5x UNL and calculated/measured creatinine clearance ≥60 ml/min)
* Measurable and/or evaluable metastatic disease

Exclusion criteria:

* Any prior palliative chemotherapy
* Neurosensory symptoms National Cancer Institute Common Toxicity Criteria for Adverse Events grade≥2

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2006-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Van Cutsem E, Boni C, Tabernero J, Massuti B, Middleton G, Dane F, Reichardt P, Pimentel FL, Cohn A, Follana P, Clemens M, Zaniboni A, Moiseyenko V, Harrison M, Richards DA, Prenen H, Pernot S, Ecstein-Fraisse E, Hitier S, Rougier P. Docetaxel plus oxaliplatin with or without fluorouracil or capecitabine in metastatic or locally recurrent gastric cancer: a randomized phase II study. Ann Oncol. 2015 Jan;26(1):149-156. doi: 10.1093/annonc/mdu496. PMID 25416687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 275 participants from 12 countries were randomized in the part I/II study. 64 participants were enrolled in Part I. 211 new participants were enrolled specifically for Part II.
Pre-assignment Details: The intent-to-treat (ITT) population, included 254 participants randomized to the optimal dose of study medication from Parts I (43) and II (211), and excluded 21 participants administered the non-optimal dose in Part I.
Groups:
- (TE) Taxotere and Eloxatin: Participants administered Docetaxel (Taxotere) 75 mg/m² as an 1-hour IV infusion on day 1 followed by Oxaliplatin (Eloxatin) 130 mg/m² as a two to six-hour IV infusion on day 1 per chemotherapy cycle.
- (TEF) Taxotere, Eloxatin and 5-fluorouracil: Participants administed with Docetaxel (Taxotere) 50 mg/m² as a 1-hour IV infusion day 1; Oxaliplatin (Eloxatin) 85 mg/m² simultaneously with folinic acid 400 mg/m² as a 2-hour IV infusion, followed by 5-FU 2400 mg/m² as a 46-hour continuous infusion day 1 per chemotherapy cycle.
- (TEX) Taxotere, Eloxatin and Xeloda: Participants administered Docetaxel (Taxotere) 50 mg/m² as a 1-hour intravenous (IV) infusion on day 1, Oxaliplatin (Eloxatin) 100 mg/m² as a two to six-hour IV infusion on day 1, Capecitabine (Xeloda) 625 mg/m2 two times a day continuously per chemotherapy cycle.
Period: Overall Study
Arm/Group | (TE) Taxotere and Eloxatin | (TEF) Taxotere, Eloxatin and 5-fluorouracil | (TEX) Taxotere, Eloxatin and Xeloda
Started | 79 | 89 | 86
Administered Non-Optimal Dose (Part I) | 10 | 11 | 0
Administered Optimal Dose (Parts I & II) | 78 | 88 | 82
Full Analysis Population (FAP) | 78 (ITT who received at least one dose of study medication) | 88 (ITT who received at least one dose of study medication) | 82 (ITT who received at least one dose of study medication)
Completed | 0 | 0 | 0
Not Completed | 79 | 89 | 86
Not completed — Adverse Event | 21 | 23 | 15
Not completed — Protocol Violation | 2 | 5 | 1
Not completed — Death | 0 | 1 | 2
Not completed — Progressive disease | 37 | 28 | 38
Not completed — Withdrew consent | 1 | 1 | 2
Not completed — Withdrawal by Subject | 11 | 20 | 12
Not completed — Surgery | 1 | 1 | 4
Not completed — Patient did not receive study medication | 1 | 1 | 4
Not completed — Clinically progressive disease | 0 | 1 | 0
Not completed — Good prognosis | 0 | 1 | 0
Not completed — Investigator/Clinical decision | 5 | 6 | 6
Not completed — Discontinued at end of study | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (TE) Taxotere and Eloxatin | (TEF) Taxotere, Eloxatin and 5-fluorouracil | (TEX) Taxotere, Eloxatin and Xeloda | Total
Number analyzed (Participants) | 79 | 89 | 86 | 254
Age Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.4) | 57.9 (11.1) | 59.0 (11.0) | 58.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 22 | 78
  Male | 51 | 61 | 64 | 176
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Oriental | 0 | 1 | 0 | 1
  Black | 1 | 0 | 0 | 1
  White | 77 | 87 | 84 | 248
  Unknown or Not Reported | 1 | 1 | 2 | 4
Karnofsky Performance Status (KPS) [Number; unit: participants]
  100% Normal, no complaints: no evidence of disease | 19 | 28 | 19 | 66
  90% Able to carry on normal activity; minor signs | 26 | 35 | 31 | 92
  80% Normal activity with effort, some signs | 31 | 24 | 33 | 88
  70% Cares for self but unable to work | 1 | 2 | 3 | 6
  <70% Requires assistance | 1 | 0 | 0 | 1
  Missing | 1 | 0 | 0 | 1
Weight loss during last 3 months [Number; unit: participants]
  less than or equal to 5% | 39 | 47 | 44 | 130
  greater than 5% | 39 | 42 | 41 | 122
  Missing | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: The number of months measured from the day of randomization to the first tumor progression according to World Health Organization (WHO) criteria evaluation of cancer response, or death from any cause.
  WHO Criteria for Progressive Disease: ≥ 25% increase in the size of at least one bidimensionally or unidimensionally measurable lesion.
Time Frame: every 8 weeks up to a maximum of 36 months
Population: 248 participants in the full analysis population (FAP).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | (TE) Taxotere and Eloxatin | (TEF) Taxotere, Eloxatin and 5-fluorouracil | (TEX) Taxotere, Eloxatin and Xeloda
Number analyzed (Participants) | 78 | 88 | 82
Months | 4.50 [3.68 to 5.32] | 7.66 [6.97 to 9.40] | 5.55 [4.30 to 6.37]

2. Secondary Outcome: Best Overall Response Rate (ORR)
Description: Percentage of partial and complete responses, according to WHO criteria:
  Complete Response: Disappearance of all known disease, determined by 2 observations not less than 4 weeks apart.
  Partial Response: Decrease by at least 50% of the diameters of all measurable lesions, determined by 2 observations not less than 4 weeks apart.
Time Frame: every 8 weeks up to a maximum of 36 months
Population: 248 participants in the full analysis population (FAP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | (TE) Taxotere and Eloxatin | (TEF) Taxotere, Eloxatin and 5-fluorouracil | (TEX) Taxotere, Eloxatin and Xeloda
Number analyzed (Participants) | 78 | 88 | 82
percentage of participants | 23.1 [14.3 to 34.0] | 46.6 [35.9 to 57.5] | 25.6 [16.6 to 36.4]

3. Secondary Outcome: Overall Survival (OS)
Description: The number of months measured from the date of randomization to the date of death due to any cause.
Time Frame: up to a maximum of 36 months
Population: 248 participants in the full analysis population (FAP).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | (TE) Taxotere and Eloxatin | (TEF) Taxotere, Eloxatin and 5-fluorouracil | (TEX) Taxotere, Eloxatin and Xeloda
Number analyzed (Participants) | 78 | 88 | 82
months | 8.97 [7.79 to 10.87] | 14.59 [11.70 to 21.78] | 11.30 [8.08 to 14.03]

ADVERSE EVENTS:
Description: 248 participants in the full analysis population (FAP) were analyzed for safety.
Arm/Group | (TE) Taxotere and Eloxatin | (TEF) Taxotere, Eloxatin and 5-fluorouracil | (TEX) Taxotere, Eloxatin and Xeloda
Serious Adverse Events (participants affected / at risk) | 35/78 | 24/88 | 36/82
Other Adverse Events (participants affected / at risk) | 75/78 | 87/88 | 77/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (TE) Taxotere and Eloxatin (N=78) | (TEF) Taxotere, Eloxatin and 5-fluorouracil (N=88) | (TEX) Taxotere, Eloxatin and Xeloda (N=82)
diarrhea (Gastrointestinal disorders) | 7 | 3 | 2
vomiting (Gastrointestinal disorders) | 2 | 3 | 3
abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
dysphagia (Gastrointestinal disorders) | 1 | 0 | 2
nausea (Gastrointestinal disorders) | 0 | 1 | 2
ascites (Gastrointestinal disorders) | 0 | 0 | 2
gastric perforation (Gastrointestinal disorders) | 0 | 1 | 1
intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
colitis (Gastrointestinal disorders) | 1 | 0 | 0
enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
hematemesis (Gastrointestinal disorders) | 0 | 0 | 1
ileus (Gastrointestinal disorders) | 0 | 1 | 0
inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0
rectal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
volvulus (Gastrointestinal disorders) | 0 | 1 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 7 | 2 | 5
anemia (Blood and lymphatic system disorders) | 2 | 0 | 1
neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
general physical health deterioration (General disorders) | 3 | 1 | 1
pyrexia (General disorders) | 2 | 1 | 0
implant site reaction (General disorders) | 0 | 0 | 2
mucosal inflammation (General disorders) | 0 | 0 | 2
performance status decreased (General disorders) | 1 | 0 | 1
asthenia (General disorders) | 0 | 0 | 1
chest pain (General disorders) | 0 | 1 | 0
device occlusion (General disorders) | 0 | 0 | 1
fatigue (General disorders) | 0 | 0 | 1
generalised edema (General disorders) | 0 | 1 | 0
device related infection (Infections and infestations) | 0 | 1 | 1
gastroenteritis (Infections and infestations) | 2 | 0 | 0
pneumonia (Infections and infestations) | 0 | 1 | 1
abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
bronchopneumonia (Infections and infestations) | 1 | 0 | 0
clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
device related sepsis (Infections and infestations) | 0 | 0 | 1
infection (Infections and infestations) | 0 | 1 | 0
neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
pelvic abscess (Infections and infestations) | 0 | 1 | 0
peritoneal abscess (Infections and infestations) | 0 | 1 | 0
sepsis (Infections and infestations) | 1 | 0 | 0
septic arthritis staphylococcal (Infections and infestations) | 1 | 0 | 0
staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
dysesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3
dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
hypovolemia (Metabolism and nutrition disorders) | 0 | 0 | 1
myocardial infarction (Cardiac disorders) | 1 | 0 | 1
cardiac failure (Cardiac disorders) | 0 | 1 | 0
cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
ataxia (Nervous system disorders) | 1 | 0 | 0
facial paresis (Nervous system disorders) | 0 | 1 | 0
headache (Nervous system disorders) | 1 | 0 | 0
peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
syncope (Nervous system disorders) | 0 | 0 | 1
deep vein thromosis (Vascular disorders) | 2 | 1 | 0
cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
investigations (Congenital, familial and genetic disorders) | 0 | 0 | 1
hemoglobin decreased (Congenital, familial and genetic disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | (TE) Taxotere and Eloxatin (N=78) | (TEF) Taxotere, Eloxatin and 5-fluorouracil (N=88) | (TEX) Taxotere, Eloxatin and Xeloda (N=82)
diarrhoea (Gastrointestinal disorders) | 48 | 59 | 53
nausea (Gastrointestinal disorders) | 45 | 52 | 43
vomiting (Gastrointestinal disorders) | 36 | 30 | 30
stomatitis (Gastrointestinal disorders) | 19 | 39 | 21
abdominal pain (Gastrointestinal disorders) | 24 | 19 | 16
constipation (Gastrointestinal disorders) | 13 | 15 | 20
abdominal pain upper (Gastrointestinal disorders) | 7 | 12 | 9
dyspepsia (Gastrointestinal disorders) | 3 | 7 | 12
dysphagia (Gastrointestinal disorders) | 6 | 5 | 10
abdominal distension (Gastrointestinal disorders) | 2 | 4 | 5
oral pain (Gastrointestinal disorders) | 4 | 0 | 1
fatigue (General disorders) | 35 | 45 | 39
asthenia (General disorders) | 21 | 22 | 16
pyrexia (General disorders) | 12 | 12 | 9
oedema peripheral (General disorders) | 8 | 10 | 12
mucosal inflammation (General disorders) | 1 | 6 | 2
oedema (General disorders) | 5 | 3 | 1
peripheral sensory neuropathy (Nervous system disorders) | 27 | 33 | 25
neuropathy peripheral (Nervous system disorders) | 12 | 19 | 19
dysgeusia (Nervous system disorders) | 5 | 23 | 12
paraesthesia (Nervous system disorders) | 11 | 16 | 6
dizziness (Nervous system disorders) | 7 | 7 | 4
headache (Nervous system disorders) | 4 | 6 | 8
dysaesthesia (Nervous system disorders) | 2 | 1 | 6
neurotoxicity (Nervous system disorders) | 4 | 3 | 0
alopecia (Skin and subcutaneous tissue disorders) | 25 | 47 | 36
nail disorder (Skin and subcutaneous tissue disorders) | 5 | 11 | 17
skin reaction (Skin and subcutaneous tissue disorders) | 4 | 5 | 13
palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 4 | 10
rash (Skin and subcutaneous tissue disorders) | 3 | 6 | 5
dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 6
decreased appetite (Metabolism and nutrition disorders) | 32 | 36 | 37
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 9
cough (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 5
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 1
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 3
hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6
back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 9
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3
hypotension (Vascular disorders) | 0 | 3 | 5
insomnia (Psychiatric disorders) | 8 | 4 | 8
anxiety (Psychiatric disorders) | 4 | 2 | 3
weight decreased (Investigations) | 5 | 7 | 8
neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 1
febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can publish the results. Prior to publication, the sponsor shall review the manuscript and can request changes, provided they do not jeopardize the accuracy and/or the scientific value of the publication. The approval is given in writing by the sponsor, not exceeding 90 days.